CLINICAL TRIAL: NCT01237873
Title: A Open-label, 52 Week, Extension to an 8-week, Double Blind, Multicenter, 6-arm, Placebo-controlled, Parallel Group Study to Evaluate the Long Term Safety of SPA100 (Aliskiren/Amlodipine)
Brief Title: Long Term Safety of SPA100 (Fixed-dose Combination of Aliskiren/Amlodipine) in Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPA100A1302
Record Dates: First submitted 2010-10-29; First posted 2010-11-10 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Essential Hypertension
Keywords: Aliskiren; Amlodipine; Essential hypertension; Long term
MeSH Terms: conditions — Essential Hypertension

ARMS (1):
- Ali/Amlo (Experimental): Aliskiren/Amlodipine 150/2.5 mg and 150/5.0 mg
  Interventions: Drug: Ali/Amlo 150/2.5 mg

INTERVENTIONS:
Drug: Ali/Amlo 150/2.5 mg — Aliskiren/Amlodipine 150/2.5 mg and 150/5.0 mg

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of the combination of aliskiren and amlodipine given to patients with essential hypertension. This study is being conducted to support registration of the fixed combination of aliskiren/amlodipine in the treatment for hypertension in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Patients that complete CSPA100A1301 study
* Patients whose blood pressure at Visit 7 of CSPA100A1301 study must be well controlled

Exclusion Criteria:

* Patients who experienced any serious adverse events considered drug related in CSPA100A1301 study
* Presence of major protocol violation in CSPA100A1301 study

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Long-term safety of the fixed-dose combination of aliskiren/ amlodipine | 52 weeks
  Measure the number patients withof AE, SAEs and analyze cahanges in safety labs.

SECONDARY OUTCOMES:
Measure the change from baseline in blood pressure effects of the combination of aliskiren/ amlodipine. | 52 weeks
  this endpoint will measure the change from baseline for mean sitting diastolic blood pressure, mean sitting systolic blood pressure, supine diastolic blood pressure, supine systolic blood pressure, standing diastolic blood pressure, and standing systolic blood pressure.
The proportion of patients achieving the blood pressure control target of <140/90 mmHg at the end of study | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Japan (12):
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Edogawa-ku, Tokyo
  - Novartis Investigative Site, Katsushika-ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Kunitachi, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shibuya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Tachikawa, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo